CLINICAL TRIAL: NCT06682780
Title: An Open-label, Dose-escalation, and Dose-expansion Phase I/II Clinical Study of Safety, Tolerability, Pharmacokinetic Profile, and Initial Efficacy of LM-2417 for Injection Alone or in Combination With Other Antitumor Agents in Patients With Advanced Solid Tumors
Brief Title: A Phase I/II Study of LM-2417 in Subjects With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM2417-01-103
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Docetaxel; toripalimab; Carboplatin; niraparib; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LM2417 Dose Escalation(Q2W/Q3W) (Experimental)
  Interventions: Drug: LM-2417
- LM-2417 combination therapy exploratory (Experimental)
  Interventions: Drug: LM-2417; Drug: Docetaxel; Drug: Toripalimab/Tirelizumab; Drug: Carboplatin; Drug: Niraparib; Drug: Lenvatinib
- LM-2417 combination expansion (Experimental)
  Interventions: Drug: LM-2417; Drug: Docetaxel; Drug: Toripalimab/Tirelizumab; Drug: Carboplatin; Drug: Niraparib; Drug: Lenvatinib

INTERVENTIONS:
Drug: LM-2417 — Q2W/Q3W,Intravenous Drip
Drug: Docetaxel — Q3W,Intravenous Drip
  Arms: LM-2417 combination expansion; LM-2417 combination therapy exploratory
Drug: Toripalimab/Tirelizumab — Q3W,Intravenous Drip
  Arms: LM-2417 combination expansion; LM-2417 combination therapy exploratory
Drug: Carboplatin — Q3W,Intravenous Drip
  Arms: LM-2417 combination expansion; LM-2417 combination therapy exploratory
Drug: Niraparib — QD,Oral Administration
  Arms: LM-2417 combination expansion; LM-2417 combination therapy exploratory
Drug: Lenvatinib — QD,Oral Administration
  Arms: LM-2417 combination expansion; LM-2417 combination therapy exploratory

SUMMARY:
This study is to assess the safety and tolerability, obtain the recommended phase 2 dose(RP2D)/or Maximum Tolerated Dose (MTD) for LM-2417 as a single agent or in combination with other anti-tumour agents in subjects with advanced solid tumours.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure.
2. Aged 18-80 years old (including boundary values) , male or female.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Life expectancy ≥ 3 months.
5. Subjects must have histological or cytological confirmation of recurrent or refractory advanced solid tumors, or currently lack or are intolerant of, standard therapy.
6. Subjects must have Archived Samples or fresh tumor tissue specimens are required for testing.
7. At least one evaluable lesion.
8. Subjects must show appropriate organ and marrow function inlaboratory examinations within 7 days prior to the first dose.
9. Women of childbearing potential (WOCBP) must agree to use highly effective methods of contraception prior to study entry, during the study and for 6 months after the last dose of study drug.
10. Subjects who can communicate well with investigators and understand and adhere to the requirements of this study.

Single-agent dose of 6mg/kg, 12mg/kg and and combined cohort：Subjects tested positive for biomarkers.

Exclusion Criteria:

1. Previously received with same target therapy.
2. Subjects has participated in any other interventional clinical trial within 28 days prior to the first dosing of LM-2417.
3. Subjects with anti-tumor treatment within 21 days prior to the first dosing of LM-2417, including radiotherapy, chemotherapy, endocrine therapy, and immunotherapy, etc.
4. Any adverse event from prior anti-tumor therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0.
5. Poorly controlled tumor-related pain.
6. Subjects with symptomatic/active central nervous system (CNS)metastases.
7. Subject who have uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
8. Subjects with known hypersensitivity to antibody therapy;
9. Subjects who take systemic corticosteroids (> 10 mg daily prednisone equivalents) for more than 7 days or other systemic immunosuppressive medications within 2 weeks prior to the first dosing of LM-2417.
10. Previous or current known autoimmune disease.
11. Subject who has interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.
12. Use of any live vaccine or live attenuated vaccines within 28 days prior to the first dosing of LM-2417.;
13. Subjects who are using therapeutic doses of anticoagulants such as heparin or vitamin K antagonists.
14. Subjects who received major surgery or interventional treatment within28 days prior to the first dosing of LM-2417.
15. Subject who have history of severe cardiovascular disease.
16. Subjects who have uncontrolled or severe illness.
17. HIV infection, active HBV or HCV infection.
18. Subjects who have other active invasive cancers, other than the one treated in this trial, within 5 years prior to screening.
19. Child-bearing potential female who have positive results in pregnancy test or are lactating.
20. Subject who have a known psychiatric diseases or disorders that may affect compliance with the trial.
21. Subject who is judged as not eligible to participate in this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-12-25 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 60 weeks
  Phase I/II
Incidence of dose-limitingtoxicity (DLT) | 60 weeks
  Phase I/II
Incidence of serious adverse event (SAE) | 60 weeks
  Phase I/II
Temperatures | 60 weeks
  Phase I/II
Pulse in BPM(Beat per Minute) | 60 weeks
  Phase I/II
Blood Pressure in mmHg | 60 weeks
  Phase I/II
Weight in Kg | 60 weeks
  Phase I/II
Height in centimeter | 60 weeks
  Phase I/II
Laboratory tests-Blood Routine examination | 60 weeks
  Phase I/II
Laboratory tests-Urine Routine test | 60 weeks
  Phase I/II
Laboratory tests-Blood biochemistry | 60 weeks
  Phase I/II
Laboratory tests- Coangulation function | 60 weeks
  Phase I/II
Echocardiography- LVEF(Left Ventricular Ejection Fraction) in percentage | 60 weeks
  Phase I/II
12-lead electrocardiogram (ECG) in HR | 60 weeks
  Phase I/II
12-lead electrocardiogram (ECG) in RR | 60 weeks
  Phase I/II
12-lead electrocardiogram (ECG) in PR | 60 weeks
  Phase I/II
12-lead electrocardiogram (ECG) in QRS | 60 weeks
  Phase I/II
12-lead electrocardiogram (ECG) in QT | 60 weeks
  Phase I/II
12-lead electrocardiogram (ECG) in QTcF | 60 weeks
  Phase I/II
ECOG(Eastern Cooperative Oncology Group) score | 60 weeks
  Phase I/II
Overall Response Rate (ORR) | 76 weeks
  Phase I/II

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax) | 112 weeks
  Phase I/II
PK Parameter:Time of Maximum Observed Concentration (Tmax) | 112 weeks
  Phase I/II
PK Parameter: Area Under the Concentration-time Curve(AUC) | 112 weeks
  Phase I/II
PK Parameter: Steady State Maximum Concentration(Cmax,ss) PK Parameter: Steady State Maximum Concentration(Cmax,ss) | 112 weeks
  Phase I/II
PK Parameter: Steady State Minimum Concentration(Cmin,ss) | 112 weeks
  Phase I/II
PK Parameter: Systemic Clearance at Steady State (CLss) | 112 weeks
  Phase I/II
PK Parameter: Accumulation Ratio (Rac) | 112 weeks
  Phase I/II
PK Parameter: Elimination Half-life (t1/2) | 112 weeks
  Phase I/II
PK Parameter: Volume of Distribution at Steady-State (Vss) | 112 weeks
  Phase I/II
PK Parameter: Degree of Fluctuation (DF) | 112 weeks
  Phase I/II
Immunogenicity of LM-2417 | 112 weeks
  Phase I/II
Biomarker correlation(NaPi2b) | 112 weeks
  Phase I/II
Duration of Response (DOR) in Month | 64 weeks
  Phase I/II
Disease control rate (DCR) in percentage | 64 weeks
  Phase I/II
progression-free survival (PFS) in Month | 64 weeks
  Phase I/II
Safety: AE/SAE (Number of participants with treatment-related adverse events as Overall survival (OS) in Month | 64 weeks
  Phase I/II
Changes of target lesions from baseline in Millimeter | 64 weeks
  Phase I/II
AE/SAE (Number of participants with treatment-related adverse events as assessed by CTCAE v5.0) Safety: AE/SAE (Number of participants with treatment-related adverse events as assessed by CTCAE v5.0) | 64 weeks
  Phase I/II

CONTACTS AND LOCATIONS:
Locations (1):
- FuDan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No